CLINICAL TRIAL: NCT01147536
Title: A Phase 2, Multicenter, Randomized, Single-Blind Study of Vitespen (HSPPC-96, Oncophage) for Immune Response Assessment Following Treatment of Patients With Resectable Renal Cell Carcinoma at Intermediate Risk of Recurrence
Brief Title: Study of Vitespen (HSPPC-96, Oncophage ®) for Immune Response Assessment in Participants With Resectable Renal Cell Carcinoma at Intermediate Risk of Recurrence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's business decision
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-100-38; NCT01073254 (obsolete NCT alias)
Record Dates: First submitted 2010-01-29; First posted 2010-06-22 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — vitespin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HSPPC-96 Vaccine (Experimental): Participants will receive up to 8 administrations of HSPPC-96 25 µg intradermally over 3 months (4 weekly doses, followed by 4 bi-weekly doses [at Weeks 14, 15, 16, 17 19, 21, 23, and 25 in Part 1a and at Weeks 1-4, 6, 8, 10, 12 in Part 1b). Participants will remain untreated with HSPPC-96 for the initial 3-month period in Part 1a for immune monitoring blood draw.
  Interventions: Biological: HSPPC-96

INTERVENTIONS:
Biological: HSPPC-96
  Other Names: HSPPC-96 (Heat Shock Protein-Peptide Complex); Prophage; Autologous Tumor-Derived HSPPC-96

SUMMARY:
The primary objective of the study is to determine whether participants exhibit a measurable immune response after multiple administrations of HSPPC-96 (heat shock protein-peptide complex 96), as assessed by enzyme linked immunosorbent spot (ELISPOT) assay.

DETAILED DESCRIPTION:
The study consists of two parts: Part 1 with Part 1a (Assessment of Immune Variation) and Part 1b (Assay Standardization), and Part 2 (Immune Monitoring Study). The study was terminated early with 12 participants enrolled only in Part 1a and Part 1b. Part 2 of the study involved randomization after 8 doses of HSSPC-96. After the 8 doses of HSSPC-96 administered in Part 2, the participants were to be randomized to the treatment extension arm or the placebo extension arm. There were no participants enrolled in Part 2 since the study was terminated early. Therefore, no randomization occurred in the conduct of this study and only a single arm was enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of histological diagnosis of renal cell carcinoma (RCC) with evidence of >= 25% clear cell carcinoma
* American joint committee on cancer tumor/node/metastasis tumor stage at intermediate risk for recurrence
* At least 8 doses of vaccine available from participant's tumor
* Life expectancy of at least 3 months
* Eastern cooperative oncology group performance status of 0 or 1
* Cardiovascular disease status of new york heart association class less than 2
* Adequate hematopoietic, renal and hepatic function
* Negative serology tests for human immunodeficiency virus (HIV), human T-cell lymphotrophic virus (HTLV-1), hepatitis B surface antigen (HBsAg), anti- hepatitis C virus antibodies (anti-HCV-Ab)
* Females must have negative pregnancy test

Exclusion Criteria:

* Evidence of metastatic or residual RCC
* Documented radiological enlarged lymph nodes
* Females who are pregnant or breastfeeding
* Use of any other investigational product from 4 weeks post-surgery
* Splenectomy performed during nephrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Lacombe, MD, FRCSC, Principal Investigator — Service d'Urologie; Centre hospitalier universitaire de Quebec - Hotel-Dieu de Quebec; Christopher G Wood, MD, FACS, Principal Investigator — M.D. Anderson Cancer Center; Ronald P Kaufman, MD, FACS, Principal Investigator — Community Care Physicians, PC; The Urological Institute of Northeastern New York
Locations (3):
- United States (2):
  - Community Care Physicians, Albany, New York
  - MD Anderson Cancer Center, Houston, Texas
- Pavillion de Recherche de Hotel Dieu, Québec, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of Part 1 (Part 1a [assessment of immune variation] and Part 2a [assay standardization]) and Part 2 (immune monitoring). Due to Business reasons, the study did not advanced to the Part 2 portion. The results presented below are for Part 1 only. Per planned analysis, data were analyzed and collected combined for Part 1a and 1b.
Groups:
- HSPPC-96 Vaccine: Participants received up to 8 administrations of HSPPC-96 (heat shock protein peptide complex-96) (Vitespen or Oncophage) 25 micrograms [µg] intradermally over 3 months (4 weekly doses, followed by 4 bi-weekly doses [at Weeks 14, 15, 16, 17 19, 21, 23, and 25 in Part 1a and at Weeks 1-4, 6, 8, 10, 12 in Part 1b). Participants remained untreated with HSPPC-96 for the initial 3-month period in Part 1a for immune monitoring blood draw.
Period: Overall Study
Arm/Group | HSPPC-96 Vaccine
Started | 12
Received at Least 1 Dose of Study Drug | 12
Completed | 9
Not Completed | 3
Not completed — Administrative study close | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug.
Groups:
- HSPPC-96 Vaccine: Participants received up to 8 administrations of HSPPC-96 25 µg intradermally over 3 months (4 weekly doses, followed by 4 bi-weekly doses [at Weeks 14, 15, 16, 17 19, 21, 23, and 25 in Part 1a and at Weeks 1-4, 6, 8, 10, 12 in Part 1b). Participants remained untreated with HSPPC-96 for the initial 3-month period in Part 1a for immune monitoring blood draw.
Arm/Group | HSPPC-96 Vaccine
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Immunological Response Using Enzyme Linked Immunosorbent Assay (ELISPOT) Assay
Description: The ELISPOT assay was not developed for this study and no immunogenicity data are available.
Time Frame: 6-7 weeks post surgery up to Week 14
Population: No Participants Provided Immunology Data. No Participants Provided Immunology Data. The ELISPOT assay was not developed for this study, and no immunogenicity data were collected for analysis.
Arm/Group | HSPPC-96 Vaccine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the date of first immune monitoring blood draw (6-7 weeks post surgery) through the end of study evaluation (12 months) or 30 days post last dose (Week 29 for Part 1a and Week 19 for Part 1b), whichever was earlier
Description: Safety population included all participants who received at least 1 dose of study drug.
Arm/Group | HSPPC-96 Vaccine
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSPPC-96 Vaccine (N=12)
Clostridium colitis (Infections and infestations) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Completed suicide (Psychiatric disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSPPC-96 Vaccine (N=12)
Anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hypercorticoidism (Endocrine disorders) | 1
Eye discharge (Eye disorders) | 1
Keratoconjuctivitis sicca (Eye disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Loose stools (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Difficulty in walking (General disorders) | 1
Fatigue (General disorders) | 3
Injection site reaction (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood pressure increased (Investigations) | 2
Blood urea increased (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Ear congestion (Ear and labyrinth disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Haemodynamic instability (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Athralgia (Musculoskeletal and connective tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Due to Business reasons, the study was terminated early and the Part 2 portion was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes